CLINICAL TRIAL: NCT05587101
Title: Optimal Diagnostic Algorithm for Neurogenic Lower Urinary Tract Symptoms in Patients With MS
Brief Title: Neurogenic Lower Urinary Tract Symptoms in Patients With Multiple Sclerosis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Koç University (Other)
Responsible Party: Sponsor
Other Study IDs: KocUrol
Record Dates: First submitted 2022-10-12; First posted 2022-10-19 (Actual); Last update posted 2022-10-19 (Actual); Status verified 2022-10

CONDITIONS: Multiple Sclerosis; Neurogenic Bladder
MeSH Terms: conditions — Multiple Sclerosis; Urinary Bladder, Neurogenic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Urodynamic Study (Filling cystometry and pressure-flow study) — Under sterile conditions and at lithotomy position, an urethral and a rectal catheter will be inserted. Bladder will be filled by sterile saline slowly. The first feeling of urine, the first sensation of urination and the sensation of severe desire to urinate will be recorded step by step. Vesical, rectal and detrusor pressures will be monitorized during these period. After the strong desire to void sensation, filling cystometry phase will be completed. Sterile saline infusion is stopped. While the patient urinates the vesical, detrusor and rectal pressures, the maximum and average urine flow rates will be recorded.
Diagnostic Test: Questionnaires — Bladder diary is an online application. Frequency, nocturia, functional bladder capacities will be reported. More than 8 urination during daytime will be recorded as overactive bladder. More than 1 interruption of sleep for urination at night is nocturia. Functional bladder capacity below 100 ml will be defined as decreased bladder capacity, while capacity over 400 ml will be reported as increased bladder capacity and compliance.
Diagnostic Test: Uroflowmetry — Uroflowmetry test consists measuring the maximum urine flow rate, the average urine flow rate, the micturiated volume and postmictional urine volume. The maximum flow rate below 12 ml/sec in males and 18 ml/sec in females will be recorded as emptying phase disorder. Postvoid residual urine volume above 150 ml is a sign of incomplete emptying of bladder.

SUMMARY:
There is no consensus in the literature upon the neurourological diagnostic algorithm of the patients with multiple sclerosis (MS). The primary aim of the study is phenotyping the patients with MS. These phenotypes might guide Neurology and Urology specialists during diagnosis and treatment. Secondary aim of this study is to define the presence and severity of urological symptoms' and disorders', involving the patients with diagnosis of MS less than 5 years into a urological follow-up and treatment process. Our study might include 4 visits (the first visit, 3rd month, 6th month and 12th month visit). Questionnaires, uroflowmetry and bladder diary might be repeated on each visit. Filling cystometry and pressure-flow study will be performed only on the first visit. All patients will receive 6 different questionnaires which aim to define the severity and presence of lower urinary tract symptoms. Bladder diary is an online application which will represent at least 3 days of frequency, urgency, incontinence episodes and the amount of fluid intake, and urination. The phenotypes would be defined after performing the first visit diagnostic tools (all of the tools are necessary during the diagnostic algorithm of neurogenic lower urinary tract symptoms). The phenotypes will be defined as: a. no symptoms with normal urodynamics, b. Lower urinary tract symptoms with normal urodynamics, c. no symptoms with abnormal urodynamics, d.lower urinary tract symptoms with abnormal urodynamics. During a follow-up period of 1 year, changes in the bladder diaries and scores in questionnaires of these groups will be compared on each visit.

ELIGIBILITY:
Inclusion Criteria:

The patients who are followed up by Department of Neurology with MS diagnosis less than 5 years

Exclusion Criteria:

1. Patients who are not eligible for completing questionnaires, bladder diaries.
2. Patients who have anatomical disorders preventing lithotomy position during urodynamic study.
3. Patients in relapsing period of MS
4. Patients who have symptoms of urinary tract infection

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patient with Multiple Sclerosis diagnosis less than 5 years
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2021-10-19 (Actual); Primary Completion 2024-01-01 (Estimated); Study Completion 2024-06-01 (Estimated)

PRIMARY OUTCOMES:
Changes in Questionnaire Scores | every 3 months
  Bladder dysfunction
Changes in Urodynamics | every 3 months
  Bladder dysfunction

CONTACTS AND LOCATIONS:
Overall Officials: Ersin Köseoğlu, Principal Investigator — Koç University
Locations (1):
- Koç University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No